CLINICAL TRIAL: NCT00623532
Title: A Randomized Interventional Study of a Cognition-Action Physical Activity and Adapted Tai-Chi in Frail Institutionalized Elderly
Brief Title: Intervention Study of Mind-Body Physical Activity in Frail Institutionalized Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association de Recherche Gerontologique (Other)
Collaborators: Conseil Régional d'Aquitaine (France) (Unknown)
Responsible Party: Isabelle Bourdel-Marchasson/ Professor (MD-PhD), Pole of Gerontology-CHU of Bordeaux/ CNRS 5536 University V Segalent Bordeaux 2
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: AGR-2006-01-Etude MARGE
Record Dates: First submitted 2008-02-15; First posted 2008-02-26 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-05

CONDITIONS: Aging; Frailty
Keywords: Tertiary prevention of disability
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CA (Experimental): Cognition and action are an inseparable whole while functioning, a new intervention based approach using familiarity based movements and non judgmental approach was labeled "cognition-action".
  Interventions: Behavioral: Mind-body exercises
- AT (Active Comparator): Adapted Tai Chi is based on Tai Chi like movements
  Interventions: Behavioral: Adapted Tai-chi
- C (No Intervention): Control

INTERVENTIONS:
Behavioral: Mind-body exercises
  Arms: CA
Behavioral: Adapted Tai-chi
  Arms: AT

SUMMARY:
Few previous studies have explored the effects of mind body approaches on health-related quality of life (HRQoL) in frail elderly. Cognition and action are an inseparable whole while functioning. A new intervention-based approach using familiarity based movements and a non-judgmental approach was labeled "cognition-action." The investigators aimed to explore the effects of two different mind-body exercise types on (HRQoL) in frail institutionalized elderly.

The investigators' main hypothesis is that adaptated physical activity in frail institutionalized elderly can improve HRQoL.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 and older
* Institutionalized
* Ability to get up alone or with technical or human help if necessary and ability to understand basic motor commands
* Have given a signed consent

Exclusion Criteria:

* Terminally ill and bedridden patients
* Unable or unwilling to sign the consent
* Have participated in a study in the past 3 month

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Actual)
Dates: Start 2006-05; Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
MOS SF-12

SECONDARY OUTCOMES:
Timed Up and Go test

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Xavier Arnozan, CHU de Bordeaux, Bordeaux, Gironde, France

REFERENCES:
- [Derived] Dechamps A, Diolez P, Thiaudiere E, Tulon A, Onifade C, Vuong T, Helmer C, Bourdel-Marchasson I. Effects of exercise programs to prevent decline in health-related quality of life in highly deconditioned institutionalized elderly persons: a randomized controlled trial. Arch Intern Med. 2010 Jan 25;170(2):162-9. doi: 10.1001/archinternmed.2009.489. PMID 20101011